CLINICAL TRIAL: NCT06591494
Title: The Efficacy of Quadruple Therapy Containing Sodium Bicarbonate as the Primary Treatment for Helicobacter Pylori Infection
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0814
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Classic quadruple therapy (Active Comparator): Esomeprazole 20 mg BID Bismuth pectin 200 mg BID Amoxicillin 1 g BID Clarithromycin 500 mg BID for 14 days
  Interventions: Drug: Classic quadruple therapy
- Quadruple therapy with sodium bicarbonate instead of bismuth (Experimental): Esomeprazole 20 mg BID Sodium bicarbonate 500 mg TID Amoxicillin 1 g BID Clarithromycin 500 mg BID for 14 days
  Interventions: Drug: Quadruple therapy with sodium bicarbonate instead of bismuth
- Quadruple therapy with sodium bicarbonate instead of clarithromycin (Experimental): Esomeprazole 20 mg BID Bismuth pectin 200 mg BID Amoxicillin 1 g BID Sodium bicarbonate 500 mg TID for 14 days
  Interventions: Drug: Quadruple therapy with sodium bicarbonate instead of clarithromycin

INTERVENTIONS:
Drug: Classic quadruple therapy — Esomeprazole 20 mg BID Bismuth pectin 200 mg BID Amoxicillin 1 g BID Clarithromycin 500 mg BID
  Arms: Classic quadruple therapy
Drug: Quadruple therapy with sodium bicarbonate instead of bismuth — Esomeprazole 20 mg BID Sodium bicarbonate 500 mg TID Amoxicillin 1 g BID Clarithromycin 500 mg BID
  Arms: Quadruple therapy with sodium bicarbonate instead of bismuth
Drug: Quadruple therapy with sodium bicarbonate instead of clarithromycin — Esomeprazole 20 mg BID Bismuth pectin 200 mg BID Amoxicillin 1 g BID Sodium bicarbonate 500 mg TID
  Arms: Quadruple therapy with sodium bicarbonate instead of clarithromycin

SUMMARY:
The goal of this clinical trial is to learn the efficacy of sodium bicarbonate-containing quadruple therapy as the primary treatment for Helicobacter pylori infection. The main questions it aims to answer are:

Can sodium bicarbonate replace bismuth or clarithromycin in the classic quadruple therapy for the primary treatment of Helicobacter pylori infection? What is the safety and cost-effectiveness of sodium bicarbonate replacing bismuth or clarithromycin in the classic quadruple therapy for the primary treatment of Helicobacter pylori infection?

Researchers will compare sodium bicarbonate replacing bismuth or clarithromycin in the classic quadruple therapy to see the efficacy of sodium bicarbonate as an alternative to bismuth or clarithromycin in the classic quadruple therapy for the primary treatment of Helicobacter pylori infection.

Participants will： Take Helicobacter pylori treatment drugs for 14 days Recheck 13C-UBT or 14C-UBT breath test 6-8 weeks after eradication treatment Incidence of adverse reactions (AEs) and patient compliance

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years, no history of eradication therapy;
* Diagnosed with Helicobacter pylori infection by one or more of the following methods: gastric mucosal histochemical staining, tissue culture, 14C-UBT, 13C-UBT and/or fecal antigen;
* Patients with warning symptoms, family history of gastric cancer or over 40 years old should undergo endoscopic examination before eradication therapy;
* Voluntarily participate in clinical trials and sign informed consent.

Exclusion Criteria:

* Use of antibiotics or bismuth within 4 weeks before enrollment, or use of acid suppressants (including H2RA, PPI or P-CAB) within 2 weeks;
* Active peptic ulcer with complications such as bleeding, perforation or obstruction;
* History of esophagectomy or gastrectomy;
* Allergy to any study drug;
* Pregnancy or lactation;
* History of alcoholism or drug abuse;
* Mental illness;
* Incapacity for civil conduct.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 855 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | 6-8 weeks after eradication treatment
  Repeat 13C-UBT or 14C-UBT breath test, negative results (<4.0‰, delta over baseline, 13C-UBT DOB; <100, DPM, 14C-UBT) indicate successful eradication. Patients are not allowed to take PPIs or P-CAB drugs 2 weeks before the breath test, and are not allowed to take antibiotics 4 weeks before the breath test.

SECONDARY OUTCOMES:
Incidence of adverse reactions (AEs) | One month after finishing with therapy
  Participants' symptoms during treatment, such as nausea, vomiting, diarrhea, rash, belching, abdominal pain, bloating, or other aggravated symptoms, were recorded and divided into three categories based on their impact on daily life: mild (transient, well tolerated), moderate (some discomfort that interferes with daily life), and severe (severe discomfort that adversely affects daily life).
Compliance of patients | One month after finishing with therapy
  Good compliance was defined as taking at least 80% of the medication.